CLINICAL TRIAL: NCT06648109
Title: Effects of Sleep Body Temperature on Body Composition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Fangfang Zeng, Associate Professor, Jinan University Guangzhou
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: JNUKY-2023-0126
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Blood Pressure Check (Hypertension Screening); Heart Rate; Aldosterone Disorder

STUDY DESIGN:
Intervention Model Description: This is a crossover controlled trial to recruit 40 people, divided into two groups of 20 subjects each using randomised grouping and named Group A and Group B. Group A will receive the sleep electric blanket intervention for a period of 7 days and Group B will serve as the control group without additional intervention, followed by a washout period of 7 days. A 1-stage baseline as well as a 3-stage follow-up including questionnaires, physical and grip strength measurements, blood index tests, and dormitory environment measurements were required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild-heat group (Experimental): Participants will be randomized into groups A and B. When the subject's group cohort undergoes the intervention phase (as opposed to the control phase), they will receive a 7-day, 8-hour intervention with an electric blanket set at +5±1°C above room temperature.
  Interventions: Device: Electric Blanket
- Non-mild-heat group (No Intervention): Participants will be randomized into groups A and B. There will be no additional sleep temperature intervention while the group is in the control period.

INTERVENTIONS:
Device: Electric Blanket — Participants were randomized to groups A and B. When the subject's group cohort went through the intervention phase (instead of the control phase), they received a 7-day, 8-hour intervention with an electric blanket +5±1°C above room temperature.
  Arms: Mild-heat group

SUMMARY:
This will be a crossover controlled trial designed to recruit 40 participants, who will be divided into two groups of 20 subjects each. The participants will be randomly assigned to either Group A or Group B. Group A will receive the sleep electric blanket intervention for a period of 7 days, while Group B will serve as the control group without any additional intervention. After the intervention period, there will be a washout period of 7 days to ensure that any effects of the intervention have subsided before the crossover.

Following the washout period, the groups will switch roles: Group B will then receive the sleep electric blanket intervention, and Group A will become the control group. This second phase will also last for 7 days, preceded and followed by the same assessment procedures as the initial phase. This design will allow for a comparison of the intervention's effects against a control period within the same group of participants, enhancing the study's internal validity.

ELIGIBILITY:
Inclusion Criteria:

- Participants aged 18-30 years, inclusive of both male and female genders.

Exclusion Criteria:

* Individuals suffering from serious diseases such as heart, liver, kidney, brain, hematopoietic, immune, thyroid, malignant tumors, etc.;
* Those with familial hereditary hypertension (both parents are hypertensive) or those diagnosed with hypertension;
* Individuals with cognitive or mental impairments that prevent the completion of the questionnaire;
* Persons with physical disabilities that hinder normal walking;
* Persons who have experienced a weight change of >3.0 kg within 1 month or >10 kg within 6 months prior to screening (as per the study in Nutrients. 2020 Oct 21;12(10):3221);
* Individuals required to take antibiotics from one week before the trial starts until its conclusion;
* Those with habitual diarrhea or who have experienced diarrhea from one week before the trial starts until its end;
* Subjects who have participated in other ambient temperature-related trials within the last 6 months;
* Individuals with extreme sleep schedules (i.e., not falling asleep between 21:00 and 2:00 a.m. the following morning, or waking up before 5:00 a.m.);
* Those with sleep latency (the time it takes to fall asleep after going to bed) greater than one hour;
* Pittsburgh Sleep Quality Index (PSQI) scores greater than 16;
* Participants who do not sign the informed consent form or are deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 1month
  Including systolic blood pressure (SBP) and diastolic blood pressure (DBP), Includes office blood pressure, home blood pressure and ambulatory blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan University Guangzhou, Guangzhou, Select A State, China

IPD SHARING:
Plan to Share IPD: Yes
The experiment will be made public upon completion with the publication of the related paper, sharing: contact the researcher for a copy.
Supporting Information: Study Protocol, ICF